CLINICAL TRIAL: NCT05409534
Title: The Effect of Backward Walking Training on Foot Biomechanics, Balance and Kinesiophobia in Elderly Individuals: A Randomized Controlled Study
Brief Title: The Effect of Backward Walking Training in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Toraman (Other)
Responsible Party: Sponsor-Investigator, Ayşe Toraman, Lecturer, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AYSE TORAMAN KARAGULMEZ
Record Dates: First submitted 2022-05-28; First posted 2022-06-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Elderly People
Keywords: balance; falls; elderly; foot
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 26 for intervention 1 (Backward Walking Exercise) group and 26 for intervention 2 (Forward Walking Home Exercise) group
Who Masked: Outcomes Assessor
Masking Description: İn this context, individuals included in the study will be assigned to the control and intervention groups respectively, randomized by an expert statistician and received in closed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backward Walking (Active Comparator): Participants who walk backward gait in the form of exercise program
  Interventions: Other: Backward Walking (Exercise group)
- Forward Walking (Active Comparator): Participants who walk forward gait in the form of home program
  Interventions: Other: Forward Walking (Control Group)

INTERVENTIONS:
Other: Backward Walking (Exercise group) — The participant will apply a maximum of 40-50 minutes of exercise, including 10 minutes of warm-up exercise, 30 minutes of backward walking training and 10 minutes of cooling-off exercise. The maximum time to do backward walking training will be 30 minutes. In the backward walking exercise, 1 set will take 5 minutes. The maximum number of sets that can be made will be 6 sets. No more than 6 sets will be made.
  Arms: Backward Walking
Other: Forward Walking (Control Group) — The participant will apply a maximum of 40-50 minutes of exercise, including 10 minutes of warm-up exercise, 30 minutes of forward walking training and 10 minutes of cooling-off exercise as the home exercise programme.
  Arms: Forward Walking

SUMMARY:
Foot problems are among the most common reasons for elderly individuals to apply to health care centers. With aging, changes occur in the appearance, biomechanics, posture and function of the foot. These changes cause deterioration in balance, increase in the risk of falling, fracture formation, limitation in mobility and activities. In recent years, backward walking seems to have become a popular treatment in rehabilitation. The walking cycle, which we start with a heel strike in our normal forward walking, starts with finger contact while walking backwards. It has been stated that this situation affects the entire plantar pressure distribution and provides a more equal distribution of plantar pressure. Therefore, gait modifications seem to affect foot biomechanics. It is not yet known how backward walking training affects foot biomechanics, balance and kinesiophobia in elderly individuals. By improving the ability to walk backwards, it may be possible to improve foot functions, increase mobility function, improve balance ability, and reduce the fear of falling and the incidence of falling. In addition, this training is easy to learn and popular, and has the advantage of being low cost. The aim of this study is to evaluate the effects of backward walking training on ankle joint position sense, foot posture and functions, lower extremity muscle strength, balance, kinesiophobia status and fall incidence in elderly individuals staying in nursing homes.

DETAILED DESCRIPTION:
The data of the research will be collected by face to face interview technique with elderly individuals living in Zonguldak Center, Kdz.Ereğli İzmirlioğlu, Devrek and Çaycuma nursing homes and meeting the inclusion criteria. In order to collect data, the "Informed Consent Form" prepared by the researcher in line with the literature will be signed by the participant and the participant's consent will be obtained. As Evaluation Methods; For socio-demographic status, Demographic Information Form, for evaluation of foot deformities and problems; Foot deformity and problems evaluation form, for disease status, Charslon Comorbidity Score for cognitive status; Standardized Mini Mental State Test for fall risk and balance assessment; Timed Get Up and Go Test for walking speed; 10 meters Forward Walk Test, 3 meters Back Walk Test, for functional capacity evaluation; Six Minute Walking Test for evaluation of dyspnea and fatigue severity; Modified Borg Scale for evaluation of foot biomechanics; Evaluation of Ankle Joint Position Sense, Foot Posture Index, Foot Function Index, for lower extremity muscle strength; Chair Sit-Up Test for fear of movement and fear of falling; Tampa Kinesiophobia Scale, International Fall Activity Scale will be used.

All tests will be carried out in the infirmary section of nursing homes, and 1 doctor, 2 nurses and equipment will be available during the practices in case of any health problems. Older adults will be evaluated by a single physical therapist with 16 years of clinical experience. All assessments will be made by the same physiotherapist. During the administration phase of the tests, a paramedic will assist in the study by standing close to the individual in case of any fall. During the application of the tests, individuals will be asked to wear the most appropriate clothes in line with their possibilities, which will make them feel comfortable, not hinder their movements. On the same day, evaluations regarding kinesiophobia and foot biomechanics will be applied to individuals. In order to minimize the effect of fatigue, tests for functional performance (timed get up and go test, 10 m forward and 3 m back walking test) will be performed on different days during the week, and the evaluations will be completed within three days.

With inspection and palpation, problems in the dominant and non-dominant feet of the individual will be recorded in the anterior, posterior and lateral view. Foot deformities such as hallux valgus, claw toe, hammer toe, mallet finger and foot problems such as calluses, dry skin and nail fungus in the participants will be evaluated and recorded.

The comorbidity score will be calculated with the "Charlson Comorbidity Index (CKI)". The scale includes 19 comorbidity scores defined according to the International Classification of Diseases 9 Clinical Modification diagnostic codes. All CKI scores are scored between 0-37. According to the results, 3 comorbidity levels are defined as low (0), moderate (1-2) and high (3+). The Standardized Mini Mental Test score will be taken into account to obtain information about the cognitive status of the participants. In this test, scores below seventeen are considered severe dementia, scores between 18-23 are considered mild dementia, and scores between 24-30 are considered normal. Universal goniometer, which is one of the valid and reliable methods used in the literature, will be used in the evaluation of ankle joint position sense of individuals. During the test, measurements will be performed by placing the pivot of the universal goniometer 1.5 cm below the lateral malleolus, the fixed arm parallel to the long axis of the fibula, and the movable arm parallel to the long axis of the 5th metatarsal, while the individuals are in the supine position, with their eyes closed to avoid visual cues. In addition, care will be taken that the goniometer does not come into contact with the individual during the measurements. Desired target angles will be determined as 10 degree dorsiflexion (DF), 10 degree plantar flexion (PF), and 20 degree PF. Individuals will be told to focus on the position of the ankle joints in space for 5 seconds by bringing their feet in the neutral position to the target position, and by repeating this process 3 times, the patient will learn this position. Then, the individual will be asked to repeat the target angle during the testing phase. Measurements will be repeated 3 times for each target angle. As a result criterion; recording the absolute value of the deviation amounts from the target angles; The average of the deviations occurring during the 3 repetitions will be taken.

Posture analysis of the foot will be made using the Foot Posture Index. Foot Posture Index; It will be evaluated according to palpation of the talus head in the posterior part of the foot, observing the inclination above and below the lateral malleolus, inversion/eversion of the calcaneus, presence of ballooning in the talonavicular joint region of the forefoot, medial longitudinal arch structure, and whether the anterior part of the foot is in abduction/adduction with respect to the posterior part of the foot. The interpretation of the test score will be done as follows; zero will indicate the neutral position of the foot, positive values will indicate the presence of pronation in the foot, and negative values will indicate the presence of supination in the foot.

The sit-stand test will be used to evaluate the lower extremity muscle strength of individuals. For the sit-stand test on a chair; A chair with a seat height of 43.18 cm, without armrests, with a straight back and a stopwatch will be used. The individual will start the test with the start command and will sit on the chair for 30 seconds. The exact number of starts during the thirty-second period will be recorded as the individual's score.

Foot Function Index is an inquiry form consisting of three sub-scales and filled by the individual himself. The Foot Function Index consists of a total of 23 questions, 9 assessing foot pain, 9 assessing disability, and 5 assessing activity limitation. Participants are asked to score all questions with a visual analog scale scaled from 0 to 10, taking into account their foot condition in the last week. Each Pain, disability, activity limitation scores and total scores for the foot will be calculated and recorded.

In the Tampa Kinesiophobia Scale, which consists of seventeen items, a 4 point likert scale was used for each item. Each item offers scoring alternatives ranging from 'strongly disagree' to 'strongly agree'. The total score is calculated after reversing the individual scores of items 4, 8, 12 and 16. Scoring ranges from 17 to 68. The cut off rate in scoring is 37, and scores below or less than 37 indicate low levels of kinesiophobia, while scores above 37 indicate high levels of kinesiophobia.

The International Falling Efficiency Scale includes 16 items scored on a 4 point scale (1=never worry, 4=very worried). The total score is scored between 16 (no anxiety) and 64 (extreme anxiety). The cut off point is 24 points to distinguish between people with a fear of falling and those without a fear of falling.

The Timed Up and Go Test is a commonly used test to evaluate balance disorders and to determine the risk of falling in the elderly. In the test, the person will be asked to get up from his chair, walk 3 meters at a safe and normal speed, turn, walk back and sit on the chair, accompanied by a stopwatch, and the time will be recorded in seconds (sec). A shorter time indicates better balance and mobility. The test starting position should be standardized. In this study, the test will be started with the individual's feet flat on the floor and the arms resting on the armrest of the chair. Three repetitions will be performed and the average of the three measurements will be recorded.

The 10-meter walking test will be used to evaluate the forward walking speed. In this test, the person walks at his/her normal speed in a pre-measured 10 meter area. Individuals will be given a warm-up distance of 3 meters to continue walking before 10 meters and 3 meters after 10 meters. The time starts when the person's foot is on the starting line of the 10-metre field and ends when he crosses the finish line. The time it takes to cover the ten meters at the person's normal speed will be recorded. The test is performed twice, and the average value is recorded with a stopwatch in m/s.

Backward walking speed will be evaluated with the 3 Meter Backward Walk Test. Colored tapes will be marked to determine the start and end line of the 3 meter area. Individuals will be asked to position their heels at the level of the horizontal band at the starting line. Individuals will be allowed to look back if they so desire. Participants will be instructed to be as fast as possible, as well as walk backwards and stop at the finish line as confidently as possible. The person administering the test will walk backwards with the participant. The test is performed once and its duration is recorded in m/s with a stopwatch.

In order to evaluate the functional exercise capacity of the individuals participating in our study, the 6-minute walking test (6MWT) will be applied to the individuals in accordance with the criteria of the American Thoracic Society. The individual will be asked to walk as much as possible at their own walking pace for six minutes on a 30-meter straight corridor. If the individual feels that he or she is unable to continue the test (such as severe dyspnea, leg pain), the individual will be told that the test will be terminated. Before starting the test, heart rate and blood pressure will be measured. At the end of the test, the assessments made before starting the test will be repeated. The walking distance of the individual will be recorded by marking the point where the test was terminated .

Modified Borg Scale will be used to evaluate the severity of dyspnea and fatigue perceived by the individual before and after the six-minute walk test. The fact that the severity of dyspnea is defined in the Modified Borg Scale makes it easier for patients to apply. This scale consists of ten items that define the severity of dyspnea according to their degrees.

For socio-demographic status, for demographic information form and disease status, Charslon Comorbidity Score will be evaluated only before treatment, all remaining assessments will be made twice, before treatment and after end of the treatment. Random assignment to intervention and control groups will be made by a statistician to avoid randomization and selection bias in the study. Participants will be included in the intervention and control groups according to random assignments after the pre-test application.Within the scope of the study, the sense of joint position of the participants will be evaluated with "Universal Goniometer", walking speed "Digital Stopwatch", walking ritms "Cherub Analog Metronome (WSM-330)", blood pressure "Sphygmomanometer (Omron M3 HEM-7155-E)".

The heart rate and blood pressure of the exercise group will be measured twice, before and after exercise. Pre-exercise heart rate and blood pressure measurement will be measured 1 cm above the elbow in the sitting position, after the individual has rested for at least 15 minutes. The post-exercise measurement will be measured from the same place as soon as the backward walking training is finished. "Sphygmomanometer (Omron M3 HEM-7155-E)" will be used for measurement of heart rate and blood pressure.Borg Scale will be used to determine exercise intensity. The perceived difficulty scale (Borg) includes numbers from 6 to 20 and corresponding difficulty expressions for these numbers.

A training program on the importance of physical activity in the elderly, prepared in line with the Turkish Physical Activity Guidelines, will be given to all participants once (in 2 sessions/30 min + 30 min) at the beginning of the study.

The heart rate and blood pressure assessments of the Backward Walking Training Group (Exercise Group) before and after each exercise will be made and the perceived difficulty levels during and after the exercise will be questioned. The Borg Scale will be explained to the individuals in the exercise group and it will be explained in detail how to indicate the level of difficulty they perceive during the exercise.

Backward walking training will consist of unimpeded gait training with or without a cane in a marked 15-meter area, on a flat surface, in optimal posture. If the individual cannot attend two sessions, these sessions will be added to the end of the 8-week exercise program and all participants will receive a total of 16 sessions. Beats per minute or bpm is the unit used to determine tempo in music. In the studies conducted in the following years, it was reported that the 60 bpm tempo in the forward and backward step tests was more easily tolerated by the elderly compared to the 120 bpm and 40 bpm tempos. As far as we know, there is no metronome tempo used during backward walking training of elderly individuals in the literature. Therefore, in our study, 50 bpm will be chosen as the starting pace, taking into account the recommended interval in the backward step tests and considering that backward walking is more difficult than forward walking. Our study is unique in that it presents backward walking training with a tempo. In order to ensure program progress in backward walking training, the tempo of the metronome will change in the range of 50-65 bpm during the 8-week training period. In the first week of the training, the tempo of the metronome will start at 50 bpm, and the tempo of the metronome will be increased by 5 bpm every 3 weeks and the program will end at 65 bpm. If the individual cannot tolerate the increase in the metronome tempo during the program progress, he/she will be able to continue his/her training at the current metronome tempo.

Before starting the backward walking training, participants will be given 10-minute warm-up exercises (breathing exercises (5 times), active ankle exercises (writing the alphabet in the sitting position, once) and standing still (2 minutes) exercise. During the movement, they will be asked to match their steps in accordance with the tempo of the metronome. While matching the tempo, the participant will be guided to alternately step with both right and left feet. Each exercise session will be individually supervised by a physiotherapist and a participant. In addition, participants will be walking backwards, standing upright. They will be encouraged to stop and look straight ahead. The training will be held in the corridor near the wall, and in case of any balance problem, the individual will be advised to "slow down and concentrate" . t will be allowed to receive support. The physiotherapist will walk a little behind the participant during the entire session, stay in close vicinity of the participant throughout the entire session and keep the participant under close surveillance. A chair will be available nearby to be used in case of need during the session. A session will last a maximum of 40-50 minutes, including warm-up exercises (10 minutes), backward walking training and cool-down exercises (10 minutes), depending on the participant's tolerance. The maximum time to climb in backward walking training will be 30 minutes. A maximum of 6 sets will be performed in five-minute periods, and no more than 6 sets will be performed. The tolerance of the participant will be taken into account in increasing the number of sets. The rest break between sets will be 2-3 minutes or as needed, and individuals will be allowed to sit while resting between sets. However, the rest breaks provided according to the discretion of the physiotherapist and the tolerance of the individuals to the activity during the gait training may be specific to the individual's needs. If individuals report that they can tolerate the increased backward walking time, the program will progress by increasing the number of sets.

After each session, the distance walked by the individuals in 5-minute periods, the number of sets and perceived difficulty levels will be recorded. In patients with complaints such as cramping, moderate to severe pain, fatigue, dizziness, weakness and palpitation during exercise, exercise training will be suspended and their continuation of the exercise program will be evaluated by re-evaluation. Individual arrangements will be made in the execution of the exercise program.

The walking training will end with cool-down exercises (10 minutes), heart rate and blood pressure measurement. As cooling exercises; the individual will be asked to perform stretching exercises for the lower extremity and waist muscles (Lumbal extensors, Hamstrings, Quadriceps, Gastro-Soleus) for 10 seconds with 4 repetitions while in a long sitting position.

To the Forward Walking Training Group(Control Group), they would apply two days a week for 8 weeks; A home program lasting 40-50 minutes in total, consisting of warm-up exercises (10 minutes), forward walking training for 30 minutes a day at the pace they feel comfortable, and cooling-down exercises (10 minutes) will be given. In addition, the participants in the control group will be visited once a week, and supervision will be given to the control group in one of every two sessions. In addition, individuals in this group will be asked to keep an activity diary, and they will be asked to write the duration of walking each week in the activity diary.

In this context, the individuals included in the research will be assigned to the control and experimental groups, respectively, and will be randomly selected by an expert statistician. The sample of the study was found at the 95% confidence interval and at the level of α= 0.05. While calculating the sample widths, since the researcher did not have any predictions about the parameters to be used in the calculation or there is no reference study in the literature that can be used to obtain the parameters, the "large effect sizes" defined by Cohen were used during the calculations. The effect size was found to be effect size = 0.80. The required sample size for the study is 52, with effect size = 0.80 for the independent sample t-test, and the minimum number of people to provide 80% test power at 95% confidence level. The sample size required for the study is effect size = 0.80 for the independent sample t-test, and the number of people who will provide the 80% test power at the 95% confidence interval is 52 in total. It was calculated as 26 people for the experimental group and 26 people for the control group. However, considering that there may be case losses, it was aimed to reach 58 people and it was planned to recruit 29 people for each group. Dependent variables of the study are foot posture index, foot function index, ankle joint position sense, kinesiophobia level, balance performance, gait speed. The independent variable is the practice of walking backwards and forwards.

The number of falls reported during the three-month period following the end of the eight-week exercise program will be learned and recorded by calling nursing homes each week. A fall will be defined as an unexpected event that results in the person lying on the ground, on the ground, or lower. When questioning the fall story, all individuals will be asked, "Have you fallen in the last 12 months?" Also it will be questioned how he/she fell if he/she fell. It will be explained that when reporting the number of falls, falls that cannot be stopped with good balance or mobility, such as trauma caused by a high-impact traffic accident, should not be included. Elderly people with a history of falling in the last 12 months will be classified as "elderly people with a history of falls" and those without a history of falling as "elderly people without a history of falls".

The study in question; According to the decision taken at the second doctoral thesis monitoring committee thesis evaluation meeting held on 22.12.2022 at 15:00, the necessity of including the six-minute walk test within the evaluation parameters in order to evaluate the effectiveness of the given backward and forward walking training on the functional capacities of the individuals was appropriate as a result of the evaluation of the first participants. seen. Accordingly, the severity of fatigue and dyspnea perceived by the individual during the implementation of the six-minute walk test will be evaluated with the Modified Borg Scale. In addition, foot deformities and problems, which are thought to be closely related to foot biomechanics, will also be evaluated observationally. The requested changes were accepted by the Health Sciences Ethics Committee with the Decision No. 23/1349 dated 03.01.2023.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age and older
* Stay in a nursing home
* Getting a score of 24 or higher on the Standardized Mini Mental State Test
* Being able to walk with a cane or without a cane
* Know how to read and write

Exclusion Criteria:

* Being vision problem that cannot be corrected with glasses or lenses
* Being hear problem that cannot be corrected with hearing aids
* Being blood pressure unsafe for exercise (>180/100 or <100/60 mmHg at rest)
* Being severe respiratory and cardiac problems (previous congestive heart failure, transient ischemic attacks)
* History of lower extremity surgery in the last six months
* Being severe orthopedic and neurological deficits that may affect walking
* History of recurrent falls (more than one fall in the last year)
* Being do exercise more than 150 minutes a week
* Participating in any exercise program in the last six months
* Three or not participating in more exercise sessions

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Balance Performance | Pre test -Post test (At the end of 8 weeks treatment)
  Timed Get Up and Go: In the test, the person will be asked to get up from his chair, walk 3 meters at a safe and normal speed, turn, walk back and sit on the chair, accompanied by a stopwatch, and the time will be recorded in seconds. Three repetitions will be performed and the average of the three measurements will be recorded. Completion of the test in a short time means better balance performance.
Lower extremity muscle strength | Pre test -Post test (At the end of 8 weeks treatment)
  Sit-Up Chair Test: The number of times the individual sits and stands in a chair during 30 seconds will be recorded as the individual's score.
Kinesiophobia | Pre test -Post test (At the end of 8 weeks treatment)
  Tampa Kinesiophobia Scale:Responses on the Tampa Kinesiophobia Scale are classified as strongly disagree, disagree, agree and strongly agree. There are two types of expressions (direct and inverse) in the scale. While these expressions are scored, those who get 1 point turn into 4, and those who get 4 points turn into 1. 4-point answers in direct statements indicate a high level of kinesiophobia. In reversed expressions, answers with a value of 1 indicate a high level of kinesiophobia, and answers with a value of 4 indicate a low level of kinesiophobia. Scores from the scale range from 17 to 68. The score obtained from the scale constitutes the individual's score that should be interpreted at the level of kinesiophobia. A high score indicates a high level of kinesiophobia.
Fear of Falling | Pre test -Post test (At the end of 8 weeks treatment)
  The International Falling Efficiency Scale: The answers given in the international fall efficiency scale are classified as (1) I am not worried at all, (2) I am a little worried, (3) I am very worried, (4) I am very worried. The total score is scored between 16 (no fear of falling) to 64 (excessive fear of falling).The cut-off point is 24 points to distinguish between people with a fear of falling and those without a fear of falling.
Forward Walking Speed | Pre test -Post test (At the end of 8 weeks treatment)
  10 meters Forward Walk Test:The time it takes to cover the ten meters at the person's normal speed will be recorded. The test is done twice and the average value is recorded in seconds. Then, 10 meters is divided by this obtained value and recorded in meters/second.
Backward Walking Speed | Pre test -Post test (At the end of 8 weeks treatment)
  3 meters Backward Walk Test:The time taken for the person to walk backwards as fast as possible will be recorded. The test is done once and its duration is recorded in seconds with a stopwatch. Then, 3 meters is divided by this obtained value and recorded in meters/second.
Foot Posture | Pre test -Post test (At the end of 8 weeks treatment)
  Foot Posture İndex: The test score is calculated by assigning values between -2 and +2 to the 6 criteria on the foot and summing the scores from all criteria.
  A test score of 0 indicates that the foot is in a neutral position. A positive test score indicates standing pronation. A negative test score indicates standing supination.
Foot Function | Pre test -Post test (At the end of 8 weeks treatment)
  Foot Function İndex:The scale consists of three subscales: pain, disability, and activity limitation. There are 23 questions in total. The participants are asked to score all questions with a visual analog scale scaled between 0-10, taking into account their foot condition in the last week. To calculate the sub-scales and the total score, the score of each item is added, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate more pain, disability, and activity limitation.
Ankle Joint Position Sense | Pre test -Post test (At the end of 8 weeks treatment)
  Individuals will be asked to bring their neutral feet to the desired target positions (10 degrees of dorsiflexion, 10 degrees of plantar flexion, 20 degrees of plantar flexion). Measurements will be repeated 3 times for each target angle. The absolute value of the deviations from the target angles will be recorded and the average of the deviations occurring during the 3 repetitions will be taken. A small amount of deviation from target angle means good Ankle Joint Position Sense.
Functional Exercise Capacity | Pre test -Post test (At the end of 8 weeks treatment)
  Six-minute walk test: The distance traveled will be measured by walking in a straight 30-meter corridor for six minutes. More distance traveled indicates better functional capacity.

SECONDARY OUTCOMES:
Cognitive status | Pre test -Post test (At the end of 8 weeks treatment)
  Standardized Mini Mental State Test: The maximum score that can be obtained from the Standardized Mini Mental State Test is 30. A score of 17 and below is considered severe dementia, a score of 18-23 is considered mild dementia, and a score of 24-30 is considered normal.
  The score obtained from the test constitutes the individual's score that should be interpreted in his cognitive state. Higher scores indicate better cognitive status.
Fall incidence | for three months after two months of treatment
  follow up by phone

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe T KARAGÜLMEZ, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Zonguldak Center, Kdz. Ereğli İzmirlioğlu, Devrek and Çaycuma Nursing Homes, Zonguldak, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since this is a doctoral thesis, it is planned to be shared after the thesis is published